CLINICAL TRIAL: NCT05165472
Title: Priming Effects of Ultra-high Frequency Quattro Pulse Transcranial Brain Stimulation Prior to Hand Motor Function Training in Children With Unilateral Spastic Cerebral Palsy
Acronym: TRAINCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRA-MAL-0034-I
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy, Spastic; Transcranial Magnetic Stimulation, Repetitive
Keywords: Unilateral Spastic Cerebral Palsy; Cortico-spinal Reorganization; Transcranial Magnetic Stimulation; Sham-controlled Trial; Intensive Hand Function Training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomized, sham-controlled, patient- and evaluator-blind, two-centre, parallel group study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Real transcranial magnetic stimulation applied
  Interventions: Other: Quadri-pulse theta burst stimulation
- Sahm-control (Sham Comparator): Sham transcranial magnetic stimulation applied
  Interventions: Other: Quadri-pulse theta burst stimulation

INTERVENTIONS:
Other: Quadri-pulse theta burst stimulation — High frequency transcranial quadri-pulse theta burst stimulation prior to hand motor function training

SUMMARY:
Unilateral spastic cerebral palsy (USCP) leads to life-long impairment with a hemiparesis of the affected side of the body. Rehabilitation efforts combine evidence based methods such as constrained induced movement therapy (CIMT) or hand-arm bimanual intensive therapy (HABIT) as well as training in daily life activities and psychological support in order to improve participation. It has been tried to enhance hand motor function trainings with non-invasive brain stimulation. However, evidence of this promising approach is limited. This might be due to a non-consideration of the individually different types of cortico-spinal projections to the paretic hand that demonstrated to be of highly relevant for the therapy of these children. Approximately one third of such patients control their paretic hands via crossed projections from the affected hemisphere (CONTRA), while one third uses ipsilateral projections from the contralesional hemisphere (IPSI). This study aims - for the first time - to enhance the effects of the training by priming the primary motor cortex (M1) of the paretic hand with a newly established high frequency quadri-pulse theta burst stimulation (qTBS) in a randomized, patient and evaluator blind, sham-controlled approach, for the first time taking the individual type of cortico-spinal reorganization (CONTRA vs IPSI) into account. This promising and neurophysiologically motivated approach is likely to ameliorate hand function in children with USCP.

ELIGIBILITY:
Inclusion Criteria:

1. Assured diagnosis of USCP.
2. Children aged 6 to 18 years with USCP
3. Dated and signed informed consent of legal guardian, informed assent from minor

Exclusion Criteria:

1. Therapy refractory epilepsy
2. Seizures within the last 2 years
3. More than 1 anti epileptic drugs
4. Implanted shunt system
5. If singular primary motor cortex cannot be identified by TMS, e.g. because of bilateral cortico-spinal reorganization or resting motor threshold above 80% maximum stimulator output (MSO)
6. Severe mental retardation
7. Psychiatric diseases
8. Pregnancy
9. Uncooperative patients

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Assisting hand assessment | 10 days
  Difference in change of logit assisting hand assessment scores between the TMS and sham-TMS group from baseline to end of 10 days intensive hand function training.

SECONDARY OUTCOMES:
Corticospinal reorganization | 1 year
  Subgroup analyses of the primary endpoint (cortico-spinal organization, age and sex) will be computed.
Assisting hand assessement - smallest detectable difference | 1 year
  Number of patients per treatment group who achieved the smallest detectable difference in logit assisting hand assessment score of 5 points at visit 12.
Assisting hand assessement - Follow up | 1 year
  Difference in the assisting hand assessment logit score between the TMS and sham-TMS group 12 months after the standardized hand motor function training.
Neuronal plasticity | 1 year
  Differences in neuronal plasticity as measured by motor evoked potentials with suprathreshold TMS single pulses between baseline and visit 12 as well as after 12 months follow-up.
Box-and-blocks test | 1 year
  Differences of Blocks transferred with the Box-and-blocks test between the TMS and sham-TMS group between baseline and visit 12 as well as after 12 months follow-up
Goal attainment scaling | 1 year
  Differences in Goal Attainment Scaling between the TMS and sham-TMS group between baseline and visit 12 as well as after 12 months follow-up.
Canadian occupational performance measure | 1 year
  Differences in the Canadian Occupational Performance Measure scale between the TMS and sham-TMS group between baseline and visit 12 as well as after 12 months follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Technical University Munich, Munich
  - Clinic for Neuropediatrics and Neurorehabilitation, Epilepsy Center for Children and Adolescents, Schön Klinik, Vogtareuth

IPD SHARING:
Plan to Share IPD: Yes
Sharing upon request planned
Supporting Information: Study Protocol, SAP
Access Criteria: The study protocol will be published in an international journal. Data will be available for other reseachers upon request.